CLINICAL TRIAL: NCT00517439
Title: A Randomized, Double-blinded Study to Evaluate the Safety and Effect on Sustained Virological Response of HCV Polymerase Inhibitor Pro-drug in Combination With PEGASYS Plus Copegus, Compared With the Currently Approved Combination of PEGASYS Plus Copegus, in Treatment-naïve Patients With Chronic he
Brief Title: A Study of Hepatitis C Virus (HCV) Polymerase Inhibitor Pro-Drug in Combination With PEGASYS Plus COPEGUS Compared With PEGASYS Plus COPEGUS in Patients With Chronic Hepatitis C Genotype 1 Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV19865
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Group 1 (Experimental): Group 1 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (1000 po bid) plus PEGASYS (180 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd).
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 2 (Experimental): Group 2 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (500 mg po bid) plus PEGASYS (180 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd).
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 3 (Experimental): Group 3 will receive HCV polymerase inhibitor pro-drug 500mg po bid plus PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd for 24 weeks; after 24 weeks, those achieving a rapid virological response (RVR) will stop all medication, and non-RVR patients will remain on triple combination for an additional 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 4 (Experimental): Group 4 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (1500 mg po bid) plus PEGASYS (90 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd).
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 5 (Experimental): Group 5 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (1000 mg po bid) plus PEGASYS (90 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd).
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 6 (Experimental): Group 6 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (500 mg po bid) plus PEGASYS (90 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd).
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO4588161
- Group 7 (Active Comparator): Standard of care (SOC)
  Interventions: Drug: Copegus; Drug: Pegasys

INTERVENTIONS:
Drug: Copegus — 1000/1200mg po daily for 24 weeks
Drug: Pegasys — 180 micrograms sc weekly for 24 weeks
  Arms: Group 1; Group 2; Group 3; Group 7
Drug: Pegasys — 90 micrograms sc weekly for 24 weeks
  Arms: Group 4; Group 5; Group 6
Drug: RO4588161 — 1000mg po bid for 24 weeks
  Arms: Group 1; Group 5
Drug: RO4588161 — 500mg po bid for 24 weeks
  Arms: Group 2; Group 3; Group 6
Drug: RO4588161 — 1500mg po bid for 24 weeks
  Arms: Group 4

SUMMARY:
This 7 arm study will determine the optimal treatment combination, based on efficacy and safety. Patients with chronic hepatitis C (CHC), genotype 1, will be randomized to one of 7 treatment groups. Groups 1, 2, 4, 5 and 6 will receive triple combination treatment with HCV polymerase inhibitor pro-drug (at doses of 500, 1000 or 1500mg po bid) plus PEGASYS (90 or 180 micrograms sc weekly) plus Copegus (1000 or 1200mg po qd) for 24 weeks, followed by 24 weeks of open label Standard of Care (PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd). Group 3 will receive HCV polymerase inhibitor pro-drug 500mg po bid plus PEGASYS 180 micrograms sc weekly plus Copegus 1000/1200mg po qd for 24 weeks; after 24 weeks, those achieving a rapid virological response (RVR) will stop all medication, and non-RVR patients will remain on triple combination for an additional 24 weeks. Group 7 will receive standard of care (SOC) for 48 weeks. There will be a 24 week period of treatment-free follow-up for all treatment groups. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* chronic hepatitis C, genotype 1;
* chronic liver disease consistent with CHC;
* compensated liver disease.

Exclusion Criteria:

* infection with any HCV genotype other than genotype 1;
* previous treatment for CHC;
* medical condition associated with chronic liver disease other than CHC;
* HIV, hepatitis A, hepatitis B infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 24 weeks post treatment end (ie weeks 48 or 72)

SECONDARY OUTCOMES:
Virological response over time | Throughout study
SVR | 12 weeks post treatment end (ie weeks 36 or 60)
Relapse rate | End of treatment (ie weeks 24 or 48)
Adverse events (AEs), laboratory parameters. | Throughout treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- United States (29):
  - Phoenix, Arizona
  - La Jolla, California
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Bradenton, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Plymouth, Minnesota
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Richmond, Virginia
- Australia (4):
  - Adelaide
  - Greenslopes
  - Melbourne
  - Sydney
- Vienna, Austria
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
- France (6):
  - Clichy
  - Créteil
  - Marseille
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Cologne
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
- Italy (3):
  - Bologna
  - Napoli
  - Torino
- Santurce, Puerto Rico
- Spain (5):
  - Badalona
  - Barcelona
  - Madrid
  - Seville
  - Valencia

REFERENCES:
- [Derived] Nelson DR, Zeuzem S, Andreone P, Ferenci P, Herring R, Jensen DM, Marcellin P, Pockros PJ, Rodriguez-Torres M, Rossaro L, Rustgi VK, Sepe T, Sulkowski M, Thomason IR, Yoshida EM, Chan A, Hill G. Balapiravir plus peginterferon alfa-2a (40KD)/ribavirin in a randomized trial of hepatitis C genotype 1 patients. Ann Hepatol. 2012 Jan-Feb;11(1):15-31. PMID 22166557